CLINICAL TRIAL: NCT05780814
Title: The Effects of Treating Insomnia on Behavioral Weight Loss Outcomes in Survivors of Breast Cancer
Acronym: COIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00376235; R01CA281220 (NIH)
Record Dates: First submitted 2023-03-09; First posted 2023-03-23 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Insomnia; Weight Gain
Keywords: women; breast cancer; weight gain; weight loss; insomnia; sleep
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders; Weight Gain; Weight Loss | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioral Therapy for Insomnia (CBT-I) (Experimental): The proposed intervention consists of 6 remotely-delivered sessions; Weeks 1, 2, 4, 6, 7, and 8, with weeks 3 and 5 being "rest weeks". Session 1 will be 60-90 mins, Session 2 will be ~60 mins, and remaining visits are ~45 mins. The investigators propose a methodological innovation for CBT-I, which involves conducting 15-minute sessions every other month during the BWL intervention. Prior to these maintenance sessions, participants in the CBT-I+BWL group will complete electronic sleep diaries for one week and interventionists will use this information in sessions to sustain and enhance long-term outcomes by using MI to reinforce application of CBT-I session content.
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Insomnia (CBT-I)
- Sleep Education Control (EDU) (Placebo Comparator): The EDU intervention will parallel the CBT-I intervention in number, format and length of all sessions, including maintenance sessions. It provides basic information about sleep and cancer, widely available to the public. EDU content does not include any individualized behavioral instructions, sleep diary monitoring during the intervention, or behavior change counseling. Content is presented didactically only.
  Interventions: Behavioral: Sleep Education Control (EDU)

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Insomnia (CBT-I) — The CBT-I intervention is a 6-session intervention spread out over 8 weeks that combines education and behavioral techniques to reduce insomnia.
  Arms: Cognitive-Behavioral Therapy for Insomnia (CBT-I)
Behavioral: Sleep Education Control (EDU) — Subjects will be instructed to read and review select publications from the American Academy of Sleep Medicine
  Arms: Sleep Education Control (EDU)

SUMMARY:
The investigators propose a randomized controlled clinical trial in 250 women with a history of early stage breast cancer who are overweight or obese with insomnia to test whether a brief, cognitive-behavioral intervention for insomnia (CBT-I) prior to behavioral weight loss (CBT-I+BWL) is superior to a sleep education control (EDU) condition followed by behavioral weight loss (EDU+BWL). The investigators will measure outcomes at baseline, 8 weeks (after completing CBT-I or EDU and prior to BWL), and at 3, 6, and 12 months.

DETAILED DESCRIPTION:
The entire study will span a 14-month period and involves one video screening visit (V1) and 4 in-person assessment visits (V2-V5) and 27 video sessions (6 for sleep intervention or sleep control and 19 for BWL). After passing an initial phone screen, participants will be scheduled for in-depth screening (V1). The investigators will complete urine samples for pregnancy and substances, administer study measures, obtain weight, height, anthropometrics and randomize at in-person visit (V2). The overall framework of the BWL intervention is social cognitive theory (increasing self-efficacy and social support) with motivational interviewing (MI) as an approach to helping participants engage in established behavior change strategies (e.g. self-monitoring, stimulus control, goal setting, feedback, etc.) aimed at reducing dietary intake and increasing physical activity (PA). Body composition will be assessed by Dual Energy X-Ray Absorptiometry (DEXA), which measures total and regional fat, lean tissue and bone mass. The investigators will conduct DEXA scans at two time points (V1 & V5).The investigators' primary endpoint is % total weight loss (TWL) at 12 months. The investigators will measure weight in light clothes without shoes, using a digital scale and height to the nearest 0.1 cm using a calibrated stadiometer, according to standardized procedures.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Histologically-confirmed Ductal Carcinoma In Situ (DCIS) or stage I-III invasive carcinoma of the breast
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Current BMI ≥ 25 kg/m2 and weight ≤ 400 lbs
* Willing to lose 10% of body weight
* Diagnosed within 10 years with histologically-confirmed DCIS or stage I-III invasive carcinoma of the breast
* Completed local therapy (i.e. surgery and radiation therapy) and any planned preoperative or adjuvant chemotherapy/immunotherapy(/HER2) human epidermal growth factor receptor 2 therapy/targeted therapy at least 3months prior to enrollment (concomitant endocrine therapy allowed)
* Completed all planned/elective surgeries >4 weeks before enrollment
* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for Insomnia disorder
* Self-reported initial sleep onset time and/or wake after sleep onset (WASO) time > 30 minutes, > 3 nights/week
* Reports sleep problems present for ≥ 3 months
* Insomnia Severity Index Score ≥ 9

Exclusion Criteria:

* Serious/uncontrolled medical or psychiatric condition likely to hinder participation in BWL or CBT-l (bipolar disorder, psychotic disorder, seizure disorders, autoimmune disease, etc.)
* Current use of medications that cause sleep disturbances or weight gain/loss. (-) Current sedative hypnotic use
* Sleep disorder other than insomnia (mild sleep apnea or moderate to severe sleep apnea successfully treated via positive airway pressure (PAP) therapy is permitted
* Currently enrolled or planning to enroll in a sleep treatment or weight loss program (agree not to enroll for the duration of the study) (-) Home sleep test Apnea/hypopnea Index (AHI) > 15
* Participants also agree not to enroll in such a program for the duration of study participation (regardless of randomization).
* History of unstable psychiatric disorder
* Self-reported suicidal ideation or severe depressive symptoms as determined by clinical assessment, triggered by score of ≥ 20 on the Center for Epidemiologic Studies Depression (CES-D)
* Lactating, pregnant or plan to become pregnant in next 14 months
* Positive urine toxicology for recreational drugs of abuse; alcohol or substance use disorder as determined by Alcohol Use Disorders Identification Test, Adapted for Use in the United States (USAUDIT294) and/or Structured Clinical Interview (SCID)
* Daily smoker/nicotine user
* Anything that, in the opinion of the investigator, would place the subject at increased risk or preclude the patient's full compliance with or completion of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned female at birth
Enrollment: 250 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Weight (pounds) | Baseline (randomization); 8 weeks post-sleep intervention (prior to BWL); and at 3, 6, and 12 months post-BWL.
  Our primary endpoint is % total weight loss (TWL) at 12 months. We will measure weight in light clothes without shoes, using a digital scale (in pounds) and height to the nearest 0.1 cm using a calibrated stadiometer, according to standardized procedures.

SECONDARY OUTCOMES:
Diet quality as assessed by Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool | Baseline (randomization); 8 weeks post-sleep intervention (prior to BWL); and at 3, 6, and 12 months post-BWL.
  Will be measured using the Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool, which follows an automated multiple-pass methodology.
Physical activity assessed by wearing and accelerometer to track movement. | Baseline (randomization); 8 weeks post-sleep intervention (prior to BWL); and at 3, 6, and 12 months post-BWL.
  Accelerometers (ActiGraph, LLC, Fort Walton Beach, FL) will be used to assess both sedentary time and moderate to vigorous physical activity.
Body composition measured through DEXA scan | Baseline and week 61
  Body composition will be assessed by dual energy x-ray absorptiometry (DEXA), which measures total and regional fat, lean tissue and bone mass

CONTACTS AND LOCATIONS:
Overall Officials: Janelle Wilder Coughlin, PHD, Principal Investigator — Johns Hopkins University; Michael Smith, PHD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Sidney Kimmel Comprehensive Cancer Center, the Avon Foundation Breast Center at Johns Hopkins, Baltimore, Maryland
  - Johns Hopkins Bayview, Baltimore, Maryland
  - Johns Hopkins Kimmel Cancer Center at Greenspring Station, Lutherville, Maryland